CLINICAL TRIAL: NCT05193643
Title: Minimally Invasive Treatment of Primary Great Saphenous Vein (GSV) Insufficiency Using High Intensity Focused Ultrasound (HIFU) Generated by Sonovein: A Single Center Prospective Feasibility Study
Brief Title: Minimally Invasive Treatment of Primary Great Saphenous Vein (GSV) Insufficiency Using High Intensity Focused Ultrasound (HIFU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-22-881
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-07

CONDITIONS: Great Saphenous Vein Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sonovein Treatment (Experimental)
  Interventions: Device: Sonovein Treatment

INTERVENTIONS:
Device: Sonovein Treatment — The Sonovein System provides High Intensity Focused Ultrasound (HIFU) ablation of soft tissue. The energy is delivered via an extra-corporeal treatment probe, which includes an imaging system. The high-energy ultrasound waves propagate through the skin and are focused on a portion of the target tissue, generating intense heat and causing local cell apoptosis and progressive tissue volume reduction over the following months in the tissue within the focal area. The process is then repeated in a stepwise fashion to destroy the targeted tissues.

SUMMARY:
This is a one-arm, open label, prospective, single-center study. Primary objective To evaluate the feasibility of HIFU for treatment of Great Saphenous Vein using assessments of patient experience and response to treatment.

Secondary objective To assess the general safety and ablation rate outcomes following HIFU treatment of GSV

ELIGIBILITY:
Inclusion Criteria:

1. Candidate for venous procedure with primary GSV insufficiency involving reflux in the segment to be treated
2. CEAP-clinical classification ≥ 2
3. Physical condition allowing ambulation after the procedure.
4. Agree to comply with the Clinical investigation plan and follow-up schedule of the study
5. Targeted tissue reachable for treatment with the device - meaning between 5mm and 24mm below the skin surface.
6. Age over 22 years at the time of enrollment.
7. No acute venous thrombosis.
8. No complete or near complete deep vein post-thrombotic disease.
9. Patient has signed and understood the written informed consent.

Exclusion criteria

1. Patient is pregnant
2. Known allergic reaction to anesthetics to be used.
3. Legally incapacitated or imprisoned patients
4. Patient's vein target not clearly visible on the ultrasound images (in B mode) at the inclusion visit.
5. Patient participating in another clinical trial involving an investigational drug or device.
6. Ankle-brachial index <7 (ABI)
7. Undergoing active anticoagulant therapy within the last 6 months
8. Diameter of the treated anatomical segment below ≤ 2mm

   -

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Technical Feasibility | 3 months
  Technical feasibility of the procedure in terms of the procedure technical success rate

SECONDARY OUTCOMES:
Ablation of venous reflux | 3 months
  - Ablation of venous reflux (as measured by Duplex ultrasound)

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Health, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No